CLINICAL TRIAL: NCT05142462
Title: Post Market Clinical Follow-up of EUROSCUP Fixe Acetabular Cup
Status: Active, not recruiting | Type: Observational
Sponsor: EUROS (Industry)
Responsible Party: Sponsor
Other Study IDs: EC-310-01-01; 2021-A01650-41 (Other: ANSM)
Record Dates: First submitted 2021-11-24; First posted 2021-12-02 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Hip Arthropathy; Hip Osteoarthritis; Hip Necrosis; Hip Fractures; Hip Dysplasia; Hip Arthritis
MeSH Terms: conditions — Osteoarthritis, Hip; Hip Fractures; Hip Dislocation | interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- EUROSCUP Fixe: 120 patients who received EUROSCUP Fixe
  Interventions: Device: Hip arthroplasty

INTERVENTIONS:
Device: Hip arthroplasty — Hip prosthesis surgical implantation

SUMMARY:
EUROSCUP Fixe is intended for use in primary and revision total hip replacement surgery.

Hip replacement is intended to provide increased patient mobility and reduce pain by replacing the damages hip joint articulation in patients where there is evidence of sufficient sound bone to seat and support the components.

As part of post market vigilance, EUROS will collect data on EUROSCUP Fixe performances and safety

DETAILED DESCRIPTION:
Post market observational study. This study is retropective and prospective, non comparative.

ELIGIBILITY:
Inclusion Criteria:

* Patient who received EUROSCUP Fixe.
* Patient informed of its participation to the study
* Patient aged between 18 and 80 years old (<80).

Exclusion Criteria:

* Patient presenting a contraindication to EUROSCUP Fixe implantation.
* Patient who refused to participate to the study
* Vulnerable subjects

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient who fulfill the criteria of eligilibilty according to the instructions for use of EUROSCUP Fixe
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2021-10-27 (Actual); Primary Completion 2022-07-29 (Actual); Study Completion 2032-07 (Estimated)

PRIMARY OUTCOMES:
Safety of EUROSCUP Fixe | 1 year
  Collect the safety of the device trought complications occurence rate

SECONDARY OUTCOMES:
Clinical performances of EUROSCUP Fixe | 1 year
  Collect the performances of the device trought clinical scores
Radiological performances of EUROSCUP Fixe | 1 year
  Collect the performances of the device trought radiological evaluation
Survival of EUROSCUP Fixe | 10 years
  Assess the survival rate of the device

CONTACTS AND LOCATIONS:
Locations (4):
- France (4):
  - Clinique Esquirol Saint Hilaire, Agen
  - Clinique de L'Atlantique, Puilboreau
  - Centre Hospitalier SECLIN, Seclin
  - Clinique St Roch, Toulon

IPD SHARING:
Plan to Share IPD: No